CLINICAL TRIAL: NCT02311556
Title: Assessment of Early Treatment Response of Brain Metastases After Gamma-Knife Radiosurgery Using Dynamic Susceptibility-weighted Contrast-enhanced Perfusion Magnetic Resonance Imaging
Brief Title: Response of Brain Metastases After Gamma-Knife Radiosurgery Using Dynamic Susceptibility-weighted Contrast-enhanced Perfusion Magnetic Resonance Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201302018
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DSC-PMR (Experimental): DSC-PMR (dynamic susceptibility-weighted contrast- enhanced perfusion magnetic resonance imaging) at baseline (screening or time of radiosurgery) and after radiosurgery
  Interventions: Device: dynamic susceptibility-weighted contrast-enhanced perfusion magnetic resonance imaging

INTERVENTIONS:
Device: dynamic susceptibility-weighted contrast-enhanced perfusion magnetic resonance imaging
  Other Names: DSC-PMR

SUMMARY:
This study is designed to evaluate whether advanced magnetic resonance imaging (MRI) techniques such as dynamic susceptibility-weighted contrast-enhanced perfusion MRI may be used to predict treatment response of brain metastasis after radiosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed brain metastases visible on brain MRI. A biopsy of the lesion is not required as long as the patient has a biopsy-proven malignancy elsewhere and a clinician deems the lesion to be metastatic.
* At least one brain metastasis must be ≥ 1cm to allow adequate quantitative imaging measurement for DSC-PMR.
* Patient must be clinically eligible for and elect to be treated with GK alone without WBRT.
* Patient must be ≥ 18 years of age.
* Patient must have Karnofsky Performance Status (KPS) of at least 60
* Patient may be part of other clinical trials (as long as no other local treatments beyond GK such as WBRT or other local therapy are indicated to the brain) or imaging studies.
* Patient or legally authorized representative must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have any medical contraindications to MRI (e.g., unsafe foreign metallic implants, incompatible pacemaker, inability to lie still for long periods, severe to end-stage kidney disease or on hemodialysis).
* Patient must not be pregnant or breastfeeding.
* Patient must not have an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2.
* Patient must not have melanoma.
* Patient must not have hemorrhagic lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Time to local progression of each treated and evaluable brain metastasis | At time of radiosurgery and after radiosurgery (approximately 1 week)
  Tumor perfusion on DSC-PMR will be used as predictor for time to local tumor progression.

SECONDARY OUTCOMES:
Radiation necrosis | Up to 1 year
  Radiation necrosis will be defined by pathology, when available. When no pathology is available, clinical diagnosis based on clinical course and management will be used.
Complete response | Up to 1 year
  Complete response = no residue enhancing lesion on MRI
Elsewhere brain failure | Up to 1 year
  Elsewhere brain failure = appearance of brain metastases outside of the prior radiosurgery region which can be diagnosed radiographically and does not required require pathological confirmation.
Clinical deterioration | Up to 1 year
  Clinical deterioration will be assessed based on the Karnofsky Performance scale (KPS).
  * 100=Normal no complaints; no evidence of disease.
  * 90=Able to carry on normal activity; minor signs or symptoms of disease.
  * 80=Normal activity with effort; some signs or symptoms of disease.
  * 70=Cares for self; unable to carry on normal activity or to do active work.
  * 60=Requires occasional assistance, but is able to care for most of his personal needs.
  * 50=Requires considerable assistance and frequent medical care.
  * 40=Disabled; requires special care and assistance.
  * 30=Severely disabled; hospital admission is indicated although death not imminent.
  * 20=Very sick; hospital admission necessary; active supportive treatment necessary.
  * 10=Moribund; fatal processes progressing rapidly.
  * 0=Dead

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu